CLINICAL TRIAL: NCT06592196
Title: A Retrospective Study on the Hepatic Safety of Statin Use in Neurology Inpatients
Brief Title: Hepatic Safety of Statin Use in Neurology Inpatients
Status: Recruiting | Type: Observational
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-154
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Statin Adverse Reaction
MeSH Terms: interventions — Coloring Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cross-sectional study and retrospective cohort study: This research was conducted in two phases. Initially, a cross-sectional study was performed to assess the correlation between statin usage prior to hospital admission and the initial state of liver enzymes among patients. Subsequently, a retrospective cohort study was undertaken, wherein patients who had not been on statins prior to admission were categorized into two groups based on their statin usage post-admission.
  Interventions: Other: stain

INTERVENTIONS:
Other: stain — This research was conducted in two phases. Initially, a cross-sectional study was performed to assess the correlation between statin usage prior to hospital admission and the initial state of liver enzymes among patients. Subsequently, a retrospective cohort study was undertaken, wherein patients who had not been on statins prior to admission were categorized into two groups based on their statin usage post-admission.

SUMMARY:
This research employs a cross-sectional study and a retrospective cohort study to analyze the liver safety of statin use among inpatients in the neurology department in China from different perspectives. The aim is to supplement evidence-based medicine and provide guidance for the clinical use of statins.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized in the Department of Neurology of Yueyang Hospital from June 2020 to February 2023.
2. Age ≥18 and ≤85 years old, both sexes.
3. Meet the diagnostic criteria of cerebrovascular disease (L1-8B0), headache disease (L1-8A8) and dizziness and vertigo (MB48) in ICD-11.

Exclusion Criteria:

1. Incomplete medical history.
2. 1 days ≤ patients with < 7 days of prior statin use.
3. Patients with malignant tumors (ICD-11 code L1-2A0, L1-2A2, L1-2B5, L1-2E6 diseases) and hematological diseases (ICD-11 code L1-3A0, L1-3B1, L1-3B8 diseases).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients admitted to the Department of Neurology at Yueyang Hospital for cerebrovascular diseases, headaches, dizziness, and vertigo from June 2020 to February 2023.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Aspartate aminotransferase(AST) | 4weeks after admission.
  The specific value of AST, whether the AST was more than 1 times the upper limit of normal (>1×ULN), and whether it was more than 3×ULN.
Alanine aminotransferase(ALT) | 4 weeks taken after admission.
  The specific value of ALT, whether the ALT was more than 1 times the upper limit of normal (>1×ULN), and whether it was more than 3×ULN.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Yueyang Integrated Medicine Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No